CLINICAL TRIAL: NCT06159478
Title: Phase II Investigator-initiated Trial of Binimetinib in Patients With BRAF Fusion-positive Low-grade Glioma or Pancreatic Cancer (Perfume)
Brief Title: Binimetinib in Patients With BRAF Fusion-positive Low-grade Glioma or Pancreatic Cancer (Perfume)
Acronym: Perfume
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH2101/MK011
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Low-grade Glioma; Pancreatic Cancer
Keywords: BRAF fusion; BRAF rearrangement; Binimetinib
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — binimetinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Binimetinib (Experimental)
  Interventions: Drug: Binimetinib 15 MG

INTERVENTIONS:
Drug: Binimetinib 15 MG — Binimetinib 45mg is orally administered twice daily.

SUMMARY:
This study is an open-label, parallel, 2-cohort, multicenter, investigator-initiated Phase 2 trial to evaluate the efficacy and safety of binimetinib in patients with advanced or recurrent low-grade glioma or pancreatic cancer harboring BRAF fusion/rearrangement.

DETAILED DESCRIPTION:
This study is an open-label, parallel, 2-cohort, multicenter, investigator-initiated Phase 2 trial. Eligible patients are with recurrent low-grade glioma (grade 1 and grade 2 tumors according to WHO classification) or advanced or recurrent pancreatic cancer harboring BRAF fusion/rearrangement. Patients receive binimetinib 45mg administered orally, twice daily.

Analyses will be performed on each of the two cohorts:

Cohort A: low-grade glioma Cohort B: pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for both cohort A and B

1. BRAF fusion or rearrangement is detected by reimbursed NGS-based cancer gene panel tests, cancer gene panel tests performed under advanced medical treatment, or clinical study (including liquid biopsy).
2. Unresectable or recurrent
3. No symptomatic brain metastasis, carcinomatous meningitis or spinal metastasis requiring surgical intervention or radiotherapy
4. No cardiac effusion, pleural effusion, or ascites requiring treatment
5. Not received anti-cancer drug within 14 days before registration, nor received other study drug (molecular targeting drug, immune therapy) within 21 days before registration
6. Not received operation under general anesthesia within 28 days before registration
7. Not received radiation therapy (including gamma knife, cyber knife) within 14 days before registration
8. Left ventricular ejection fraction >= 50% by echocardiography or MUGA (multigated acquisition scan) within 28 days before registration
9. Having all laboratory tests performed within 14 days before registration and the values are within the following range. Patients should not receive administration of G-CSF and/or blood transfusion within 14 days before the blood collection (1) Absolute neutrophil count >= 1.500/mm3 (2) Platelet count >= 10.0 X 10(4))/mm3 (3) Hemoglobin >= 8.0 g/dL (4) Total bilirubin <= 1.5 g/dL (5) Aspartate aminotransferase (AST) <= 100 U/L (6) Alanine aminotransferase (ALT) <= 100 U/L (7) Serum creatinine <= 1.5 mg/dL
10. Patients who are able to swallow orally administered medication.
11. Consent to at least 30 days of contraception and limited egg donation (including egg retrieval for future egg transfer) after last administration of study drug for child-bearing status women. Consent to 90 days of contraception and limited sperm donation after last administration of study drug for men.
12. Written informed consent (When registering patient under 18, a signed consent form must be obtained from both the patient and the parent or legal guardian.)

    Cohort A
13. Histopathologically diagnosed as low-grade glioma, based on WHO classification of 2007, 2016 and 2021. The grade is WHO grade 1 or 2.
14. Age at the time of registration is 12 years or older (When registering a patient under 18, a signed consent form must be obtained from both the patient and the parent or legal guardian), and patients who are 12-17 years old have to be 40 kg or over in body weight. There is no limitation in body weight for patients who are 18 years or older.
15. Lansky Performance Status (LPS) >= 70 for patients 12-15 years old Karnofsky Performance Status (KPS) >= 70 for patients 16 years or older
16. Having measurable disease within 28 days before registration
17. Patients suffice the following. (1) Having adequate initial treatment depending on the primary central nervous tumor including surgery if recommended treatment is available. (2) Neurologically stable.

(3) Multiple lesion or dissemination is not detected with MRI at the registration.

18) Not increased steroid for low-grade glioma within 14 days before registration and the dosage of steroid in equivalent to 50 mg prednisolone or less.

Cohort B 19) Histopathologically diagnosed as pancreatic cancer (histologically not specified).

20) Having progression after at least one regimen of chemotherapy excluding adjuvant therapy.

21) Age at the time of registration is 18 years or older. 22) Performance Status (ECOG) is 0 or 1 23) Having measurable disease within 28 days before registration detected by enhanced CT (Head, chest, abdominal, pelvic: under 5 mm in slice)

Exclusion Criteria:

1. Active double primary cancer (but not [1]-[3]): [1] completely resected following cancers: basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, superficial bladder cancer, [2] gastrointestinal cancer curatively resected with ESD or EMR, and [3] other cancers with no recurrence for more than 5 years.
2. Patients with symptomatic congestive heart failure of NYHA class II-IV or arrythmia (over grade 2) occurring in less than 6 months before registration.
3. Patients with myocardial infarction or unstable angina occurring in less than 6 months before registration.
4. Patients with corrected QT interval (QTcF) > 480 ms in ECG performed within 14 days before enrollment.
5. Patients with infections requiring systemic treatment.
6. Patients with uncontrolled hypertension (systolic blood pressure: over 150 mmHg or diastolic blood pressure: over 100 mmHg).
7. Patients with history or findings of retinal vein occlusion (RVO) or having RVO risk factor (unstable glaucoma, ocular hypertension, hyperviscosity syndrome, hypercoagulability syndrome, etc.)
8. Patients with history or complication of retinal degenerative disease other than RVO (central serous chorioretinopathy, retinal detachment, age-related macular degeneration, etc.)
9. Patients with uncontrolled diabetes mellitis.
10. Patients with venous thrombus (transient ischemic attack, stroke, massive deep vein thrombosis, pulmonary embolism, etc.) occurring in less than 3 months
11. Patients who have neuromuscular disease with CK elevation (inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy, etc.).
12. Prior treatment with MEK inhibitors.
13. Previous severe hypersensitive reaction to ingredient including binimetinib.
14. Patients who are positive for either HIV antibody, HBs antigen, or HCV-RNA.
15. Negative for HBs antigen, positive for HBs antibody or HBc antibody, and positive for HBV-DNA assay. (If it is less than or equal to the detection sensitivity, patients are not excluded)
16. Patients with concomitant diseases that affect gastrointestinal function.
17. Women who are pregnant, breastfeeding and need to continue breastfeeding in the future, and women who may be pregnant.
18. Patients with psychiatric diseases or psychological symptoms interfering with participation in the trial.
19. Patients who are deemed inappropriate for participation in the trial by the principal investigator or sub-investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (centrally assessed) | Baseline up to 4 years
  Overall response rate (ORR) defined as the combined incidence of complete response (CR) and PR, within cohort A FAS, cohort B FAS, and confirmed no less than 4 weeks after the criteria for response are first met, based on RECIST v1.1. ORR will be confirmed by independent blinded central review assessment.

SECONDARY OUTCOMES:
Overall response rate (investigator assessed by RECIST) | Baseline up to 4 years
  Overall response rate (ORR) defined as the combined incidence of complete response (CR) and PR, within cohort A FAS, cohort B FAS, and confirmed no less than 4 weeks after the criteria for response are first met, based on RECIST v1.1. ORR will be performed by investigator assessment.
Overall response rate (investigator assessed by RANO) | Baseline up to 4 years
  Overall response rate (ORR) defined as the combined incidence of complete response (CR) and PR, within cohort A FAS, and confirmed no less than 4 weeks after the criteria for response are first met, based on Response Assessment in Neuro-Oncology (RANO) criteria. ORR will be confirmed by local site investigator assessment.
Overall response rate including minor response(investigator assessed by RANO) | Baseline up to 4 years
  Overall response rate (ORR) defined as the combined incidence of complete response (CR) PR and SD, within cohort A FAS, and confirmed no less than 4 weeks after the criteria for response are first met, based on Response Assessment in Neuro-Oncology (RANO) criteria. ORR will be confirmed by local site investigator assessment.
Progression-free survival | Baseline up to 4 years
  Progression-free survival (PFS) defined as the time from the date of enrollment to the date of the first documentation of objective progression of disease (PD), clinically diagnosed symptomatic deterioration, or death due to any cause in the absence of documented PD, whichever occurs first within cohort A FAS and cohort B FAS.
Overall survival | Baseline up to 4 years
  Overall survival (OS) defined as the time from date of enrollment to date of death due to any cause within cohort A FAS and cohort B FAS.
Disease control rate | Baseline up to 4 years
  Disease control rate (DCR) defined as the percentage of patients with a confirmed complete response (CR), partial response (PR) or stable disease (SD) as the best overall according to RECIST version 1.1 within cohort A FAS and cohort B FAS.
Duration of response | Baseline up to 4 years
  Duration of Response (DOR) defined as the time from the date of first documentation of CR or PR to the date of first documentation of disease progression or date of death from any cause, whichever occurs first within cohort A FAS and cohort B FAS.
Adverse event rate | Baseline up to 4 years
  Defined as the percentage of patients who experienced each adverse event. The severity of AEs were evaluated by the investigator according to Japan Clinical Oncology Group (JCOG) Japanese translation of the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0-JCOG) within cohort A FAS and cohort B FAS.

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku university Hospital, Sendai, Miyagi
  - National Cancer Center Japan, Chuo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: No